CLINICAL TRIAL: NCT00767780
Title: The Effect of a New Biomechanical Device
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 141/08
Record Dates: First submitted 2008-10-02; First posted 2008-10-07 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Osteoarthritis; Joint Replacement; Fractures
MeSH Terms: conditions — Osteoarthritis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 3: Patients suffering from ankle fractures and instability
  Interventions: Device: APOS biomechanical gait system
- 4: Patients suffering from hip osteoarthritis
  Interventions: Device: APOS biomechanical gait system
- 5: Patients who underwent total knee replacement or total hip replacement
  Interventions: Device: APOS biomechanical gait system
- 1: Patients suffering from bilateral knee osteoarthritis
  Interventions: Device: APOS biomechanical gait system
- 2: Patients suffering fron non specific low back pain
  Interventions: Device: APOS biomechanical gait system

INTERVENTIONS:
Device: APOS biomechanical gait system — a biomechanical device including 2 hemispheric biomechanical elements attached to a platform in a form of a shoe. the biomechanical device is calibrated to each patient by a physiotherapist specialized with the treatment methodology. patient are instructed to walk indoor with the device. time of exercise is gradually increase

SUMMARY:
The purpose of this study is to examine (retrospectively) the effect of a new biomechanical device on gait patterns of patients suffering from musculoskeletal disorders. The analysis is conducted on an existing database of the therapy center.

DETAILED DESCRIPTION:
Patients treated in the therapy center undergo a computerized gait test and complete several pain and function questionnaires at fixed time point. We examined the effect of the treatment on the level of pain, function and quality of life as well as on the gait patterns of these patients. Measurements were taken at baseline, after 3 months, and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* knee\hip OA
* knee\hip joint replacement
* ankle fractures\instability
* NSLBP

Exclusion Criteria:

* neurological disorders
* lack of balance (2 falls in the last year)
* incapable to complete a questionnaire

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from one of the following conditions: knee\hip OA, knee\hip joint replacement, ankle fractures\instability, NSLBP
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Gait spatio-temporal parameters

SECONDARY OUTCOMES:
WOMAC, SF-36, Oswestry and FAOS questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Debbi, MD, Study Director — Assaf Harophe Medical Center
Locations (1):
- APOS Medical and Sport Thechnologies LTD, Herzliya, Israel

REFERENCES:
- [Derived] Atoun E, Mor A, Segal G, Debi R, Grinberg D, Benedict Y, Rozen N, Beer Y, Elbaz A. A non-invasive, home-based biomechanical therapy for patients with spontaneous osteonecrosis of the knee. J Orthop Surg Res. 2016 Nov 14;11(1):139. doi: 10.1186/s13018-016-0472-0. PMID 27842560
- [Derived] Herman A, Chechik O, Segal G, Kosashvili Y, Lador R, Salai M, Mor A, Elbaz A, Haim A. The correlation between radiographic knee OA and clinical symptoms--do we know everything? Clin Rheumatol. 2015 Nov;34(11):1955-60. doi: 10.1007/s10067-015-2871-8. Epub 2015 Jan 22. PMID 25604319
- [Derived] Elbaz A, Beer Y, Rath E, Morag G, Segal G, Debbi EM, Wasser D, Mor A, Debi R. A unique foot-worn device for patients with degenerative meniscal tear. Knee Surg Sports Traumatol Arthrosc. 2013 Feb;21(2):380-7. doi: 10.1007/s00167-012-2026-2. Epub 2012 May 4. PMID 22555568
- [Derived] Debi R, Mor A, Segal G, Debbi EM, Cohen MS, Igolnikov I, Bar Ziv Y, Benkovich V, Bernfeld B, Rozen N, Elbaz A. Differences in gait pattern parameters between medial and anterior knee pain in patients with osteoarthritis of the knee. Clin Biomech (Bristol). 2012 Jul;27(6):584-7. doi: 10.1016/j.clinbiomech.2012.02.002. Epub 2012 Mar 9. PMID 22406298
- [Derived] Elbaz A, Debbi EM, Segal G, Haim A, Halperin N, Agar G, Mor A, Debi R. Sex and body mass index correlate with Western Ontario and McMaster Universities Osteoarthritis Index and quality of life scores in knee osteoarthritis. Arch Phys Med Rehabil. 2011 Oct;92(10):1618-23. doi: 10.1016/j.apmr.2011.05.009. Epub 2011 Aug 12. PMID 21839981
- [Derived] Elbaz A, Mor A, Segal G, Debbi E, Haim A, Halperin N, Debi R. APOS therapy improves clinical measurements and gait in patients with knee osteoarthritis. Clin Biomech (Bristol). 2010 Nov;25(9):920-5. doi: 10.1016/j.clinbiomech.2010.06.017. Epub 2010 Jul 16. PMID 20637534
- [Derived] Elbaz A, Mirovsky Y, Mor A, Enosh S, Debbi E, Segal G, Barzilay Y, Debi R. A novel biomechanical device improves gait pattern in patient with chronic nonspecific low back pain. Spine (Phila Pa 1976). 2009 Jul 1;34(15):E507-12. doi: 10.1097/BRS.0b013e3181a98d3f. PMID 19564755